CLINICAL TRIAL: NCT02819310
Title: An Open Label Study of Chronic Use of BLI400 Laxative in Constipated Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI400-303
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Constipation; Chronic Idiopathic Constipation; CIC
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLI400 Laxative (Experimental): BLI400 Laxative
  Interventions: Drug: BLI400 Laxative

INTERVENTIONS:
Drug: BLI400 Laxative — oral laxative

SUMMARY:
The objective of this study is to evaluate the safety of chronic use of BLI400 laxative in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age
2. Constipated, defined by the following adapted ROME II definition:

   * Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for at least 12 weeks (which need not be consecutive) in the preceding 12 months:
   * Straining during > 25% of defecations
   * Lumpy or hard stools in > 25% of defecations
   * Sensation of incomplete evacuation for > 25% of defecations
3. If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse)
4. Negative urine pregnancy test at screening, if applicable
5. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Report loose (mushy) or water stools in the absence of laxative use for more than 25% of BMs during the 12 weeks before Visit 1
2. Meet the Rome II criteria for Irritable Bowel Syndrome
3. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
4. Subjects who have had major surgery 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
5. Subjects with hypothyroidism that is being treated and for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of Visit 1
6. Subjects taking laxatives, enemas or prokinetic agents that refuse to discontinue these treatments from Visit 1 until after completion of Visit 6
7. Subjects who are pregnant or lactating, or intend to become pregnant during the study
8. Subjects of childbearing potential who refuse a pregnancy test
9. Subjects who are allergic to any BLI400 component
10. Subjects taking narcotic analgesics or other medications known to cause constipation.
11. Subjects with clinically significant cardiac abnormalities identified at the Visit 1 ECG
12. Subjects with clinically significant laboratory abnormalities, deemed as a potential safety issue by the Investigator, may be discontinued at the Investigator's discretion.
13. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
14. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
15. Subjects with an active history of drug or alcohol abuse
16. Subjects have been hospitalized for a psychiatric condition or have made a suicide attempt during the 2 years before Visit 1
17. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (24):
- United States (24):
  - Braintree Research Site 14, Corona, California
  - Braintree Research Site 13, Brandon, Florida
  - Braintree Research Site 3, Brandon, Florida
  - Braintree Research Site 18, Hialeah, Florida
  - Braintree Research Site 19, Hialeah, Florida
  - Braintree Research Site 4, Miami, Florida
  - Braintree Research Site 5, Miami, Florida
  - Braintree Research Site 16, Miami, Florida
  - Braintree Research Site 8, Miami Lakes, Florida
  - Braintree Research Site 17, Palmetto Bay, Florida
  - Braintree Research Site 12, St. Petersburg, Florida
  - Braintree Research Site 2, West Palm Beach, Florida
  - Braintree Research Site 24, Owensboro, Kentucky
  - Braintree Research Site 15, Lake Charles, Louisiana
  - Braintree Research Site 25, Las Vegas, Nevada
  - Braintree Research Site 21, Fayetteville, North Carolina
  - Braintree Research Site 6, Cincinnati, Ohio
  - Braintree Research Site 11, Chattanooga, Tennessee
  - Braintree Research Site 22, Memphis, Tennessee
  - Braintree Research Site 10, Nashville, Tennessee
  - Braintree Research Site 20, Carrollton, Texas
  - Braintree Research Site 23, Houston, Texas
  - Braintree Research Site 1, Plano, Texas
  - Braintree Research Site 7, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI400 Laxative
Started | 330
Completed | 221
Not Completed | 109
Not completed — Withdrawal by Subject | 37
Not completed — Lost to Follow-up | 16
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 8
Not completed — Protocol Violation | 30

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | BLI400 Laxative
Number analyzed (Participants) | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 133
  Not Hispanic or Latino | 172
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 91
  White | 205
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 305

OUTCOME MEASURES:

1. Primary Outcome: % of Subjects With Treatment Emergent Adverse Events
Description: % of subjects experiencing a treatment emergent adverse event during the 12 month treatment period
Time Frame: 12 months
Population: FDA agreed upon Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BLI400 Laxative
Number analyzed (Participants) | 305
Participants | 108

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | BLI400 Laxative
All-Cause Mortality (participants affected / at risk) | 0/305
Serious Adverse Events (participants affected / at risk) | 2/305
Other Adverse Events (participants affected / at risk) | 34/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 Laxative (N=305)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (305)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI400 Laxative (N=305)
Diarrhea (Gastrointestinal disorders) | 23 (23)
Flatulence (Gastrointestinal disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02819310/Prot_SAP_000.pdf